CLINICAL TRIAL: NCT01928836
Title: Multicenter Study for Risk Stratification of Patients Presenting With Symptoms Related to Lung Cancer Using the Lung Cancer Biomarker Panel (LCBP) in China
Brief Title: Risk Stratification of Patients Using the Lung Cancer Biomarker Panel in China
Acronym: LCBP
Status: Completed | Type: Observational
Sponsor: Bai Chunxue (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Peking Union Medical College Hospital (Other); Nanjing PLA General Hospital (Other); Third Military Medical University (Other); First Affiliated Hospital of Zhejiang University (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Bai Chunxue, Director, Chinese Alliance Against Lung Cancer
Organization: Chinese Alliance Against Lung Cancer (Other)
Other Study IDs: CAALC-001-LCBP
Record Dates: First submitted 2013-08-20; First posted 2013-08-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Lung Neoplasms
Keywords: Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Biological Markers; ROC Curve; Delayed Diagnosis
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — 10mL blood sample of the patient will be tested for cancer biomarkers, biochemical detection and cardiovascular disease biomarkers, etc.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-suspected lung cancer group: 1. Aged 40 to 75 years;
  2. Male smoker (≥400 cig/year), female smoker or non-smoker;
  3. Visible lung nodule lesion in the chest (based on local CT result);
  4. Without the indication of biopsy (bronchoscope or percutaneous transthoracic) or surgery.
- Suspected lung cancer group: 1. Aged 40 to 75 years;
  2. Male smoker (≥400 cig/year), female smoker or non-smoker;
  3. Visible lung cancer lesion in the chest (based on local CT result);
  4. With the indication of biopsy (bronchoscope or percutaneous transthoracic) or surgery.

SUMMARY:
The purpose of this study is to verify clinical utility of a simple blood test comprising of four protein- based markers for risk stratification of patients presenting symptoms related to lung cancer.

DETAILED DESCRIPTION:
The study is a multicenter, prospective case-control research. Totally 1,200 cases will be collected in the hospitals, with 600 cases in control group, which are not suspected as lung cancer from chest CT, and other 600 in suspected group. When inclusion into the two groups, clinical information and 10mL blood sample of the patient will be recorded and tested for cancer biomarkers, biochemical detection and cardiovascular disease biomarkers, etc. The correlation between cancer biomarker panel, CT scan result and clinical pathological diagnosis will be investigated through cases follow up. The sample size estimated above was set up according to sensitivity and specificity of biomarkers in pre-study, based on lung cancer incidence of the population. To compare the diagnostic accuracy among different cancer biomarkers through T-test, Mann-Whitney U and receiver operating characteristic (ROC) curve with SPSS 15.0 software. In statistic analysis, 0.05 is set as the p value for significance. Effectiveness of the four biomarkers panel in lung cancer diagnoses and staging will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Non-suspected lung cancer group (600 cases)

  1. Aged 40 to 75 years;
  2. Male smoker (≥400 cig/year), female smoker or non-smoker;
  3. Visible lung nodule lesion in the chest (based on local CT result);
  4. Without the indication of biopsy (bronchoscope or percutaneous transthoracic) or surgery.
* Suspected lung cancer group (600 cases)

  1. Aged 40 to 75 years;
  2. Male smoker (≥400 cig/year), female smoker or non-smoker;
  3. Visible lung cancer lesion in the chest (based on local CT result);
  4. With the indication of biopsy (bronchoscope or percutaneous transthoracic) or surgery.

Exclusion Criteria:

* Histopathological diagnosis result is unavailable, including patients only have cytology results of pleural effusion;
* Already treated by chemotherapy or surgery

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Totally 1,200 cases will be collected in the hospitals, with 600 cases in control group, which are not suspected as lung cancer from chest CT, and other 600 in suspected group.
Sampling Method: Non-Probability Sample
Enrollment: 764 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence rate of lung cancer | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chunxue Bai, Prof., Principal Investigator — Chinese Alliance Against Lung Cancer
Locations (6):
- China (6):
  - Peking Union Medical College Hospital, Beijing
  - Third Military Medical University, Chongqing
  - First Affiliated Hospital of Zhejiang University, Hangzhou
  - Nanjing PLA General Hospital, Nanjing
  - Shanghai Zhongshan Hospital, Shanghai
  - Henan Provincial Hospital, Zhengzhou

REFERENCES:
- [Derived] Yang D, Zhang X, Powell CA, Ni J, Wang B, Zhang J, Zhang Y, Wang L, Xu Z, Zhang L, Wu G, Song Y, Tian W, Hu JA, Zhang Y, Hu J, Hong Q, Song Y, Zhou J, Bai C. Probability of cancer in high-risk patients predicted by the protein-based lung cancer biomarker panel in China: LCBP study. Cancer. 2018 Jan 15;124(2):262-270. doi: 10.1002/cncr.31020. Epub 2017 Sep 20. PMID 28940455
- [Derived] Yang D, Zhou J, Zeng T, Yang Z, Wang X, Hu J, Song Y, Chen L, Peer D, Wang X, Bai C. Serum chemokine network correlates with chemotherapy in non-small cell lung cancer. Cancer Lett. 2015 Aug 28;365(1):57-67. doi: 10.1016/j.canlet.2015.05.001. Epub 2015 May 11. PMID 25976768